CLINICAL TRIAL: NCT07302074
Title: Understanding of Rare Inflammatory Arthritis in Comparison to Classical Inflammatory Arthritis : Tissular Observations and Immune Infiltrate Characterization : the UTOPIC Project
Acronym: UTOPIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 29BRC24.037
Record Dates: First submitted 2025-11-28; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Inflammatory Arthritis; Rare Auto-immune Diseases; Immune Checkpoint Inhibitor Related Inflamamtory Arthritis
Keywords: immune checkpoint inhibitor related inflamamtory arthritis; Inflammatory arthritis; rare auto-immune diseases; connective tissue disease
MeSH Terms: conditions — Arthritis; Connective Tissue Diseases | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Arthritis or bursitis occurring in the context of a rare MIS or drug-induced toxicity."
  Interventions: Procedure: Biopsy
- Arthritis or bursitis (Other)
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — "A synovial biopsy will be carried out as recommended

SUMMARY:
The pathophysiology of certain inflammatory arthritides remains poorly understood, particularly when associated with rare systemic autoimmune diseases such as systemic sclerosis (SSc), or when emerging in the context of immune-related adverse events from cancer immunotherapies. These immunotherapy-induced arthritides represent a new and increasingly encountered clinical entity in rheumatology. A deeper understanding of the mechanisms underlying joint inflammation in these settings is essential for identifying specific therapeutic targets, especially given the limitations of current treatment options and the risks associated with broad immunosuppressive strategies such as prolonged corticosteroid use, which may impair anti-tumor immune responses.

Synovial biopsy analysis provides a powerful tool for dissecting the cellular and molecular components of joint inflammation, including immune cell infiltration, cytokine profiles, and cell-cell interactions. Advances in high-dimensional techniques such as multiplex immunofluorescence and mass cytometry now allow for the identification and spatial localization of numerous protein markers at the subcellular level. Additionally, spatial transcriptomics offers complementary insight into gene expression profiles within the tissue microenvironment, providing a comprehensive understanding of inflammatory processes.

The investigators propose a prospective, proof-of-concept study to characterize and compare rare and emerging inflammatory arthritides-including those linked to SSc and immunotherapy-related immune toxicity-with classical inflammatory rheumatic diseases such as rheumatoid arthritis (RA), psoriatic arthritis (PsA), spondyloarthritis (SpA), polymyalgia rheumatica (PMR), and reactive arthritis. Through detailed immunological and molecular profiling, this study aims to identify disease-specific signatures and novel therapeutic targets. These findings could pave the way for precision medicine approaches and inform the development of targeted therapies in both rare and common forms of inflammatory arthritis.

ELIGIBILITY:
Inclusion Criteria:

* For all participants:

  * Signed consent form
  * Patients over 18 years old
  * Affiliated with a social security scheme
* For cases:

  * Referred for arthritis or bursitis occurring in the context of a rare systemic autoimmune disease (SAID) or drug-induced toxicity.
  * Presenting at least one clinical arthritis with synovial thickening confirmed by ultrasound (grade ≥2 in B-mode) and Doppler inflammation of grade ≥1, or synovial thickening ≥B2 associated with joint effusion.

For bursitis: thickening ≥2mm of at least one periarticular bursa on ultrasound associated with Doppler inflammation of grade ≥1, or synovial thickening ≥2mm associated with joint effusion, with clinical evidence of inflammatory involvement.

*For the control group:

For arthritis:

* Presenting clinical arthritis with synovial thickening confirmed by ultrasound (grade ≥2 in B-mode (B2)) and Doppler inflammation of grade ≥1, or synovial thickening ≥B2 associated with joint effusion.
* Diagnosed, according to disease-specific classification criteria, with either rheumatoid arthritis (according to ACR/EULAR 2010 criteria), axial or peripheral spondyloarthritis (according to ASAS 2009 criteria), psoriatic arthritis (according to CASPAR criteria), or reactive arthritis based on clinician assessment.

For bursitis:

* Thickening ≥2mm of at least one periarticular bursa on ultrasound associated with Doppler inflammation of grade ≥1, or synovial thickening ≥2mm associated with joint effusion.
* Meeting the ACR/EULAR 2012 criteria for polymyalgia rheumatica.

Exclusion Criteria:

* For all participants:

  * Patients under protective measures or unable to consent
  * Pregnant or breastfeeding women
  * Anticoagulant treatment: vitamin K antagonists (Coumadin, fluindione), direct oral anticoagulants (Eliquis, Pradaxa, Rivaroxaban), heparins at curative doses
  * Contraindication to local procedure: lymphedema near the joint, chronic wound at the site of the joint, joint prosthesis on the affected joint, corticosteroid infiltration less than 3 months ago at the same site
  * History of treatment with biotherapy or targeted therapy (JAK inhibitors) within the last 3 months, or within the last 6 months if treated with Rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
characterize the inflammatory infiltrate in synovial biopsies | Day 1
  Establishment of a biobank to characterize the inflammatory infiltrate in synovial biopsies from arthritis or bursitis occurring in the context of rare systemic autoimmune diseases (SAIDs) or immune-mediated drug toxicities, and to compare it with the infiltrate in the synovium of arthritis/bursitis associated with common inflammatory rheumatic conditions frequently encountered in rheumatology.

SECONDARY OUTCOMES:
Study of the cytokine environment | day 1
  Study of the cytokine environment within synovial biopsies from arthritis/bursitis occurring in the context of rare autoimmune/inflammatory syndromes or drug toxicity
Study of the cytokine environment | day 1
  Study of the cytokine environment within synovial biopsies fromarthritis/bursitis arising in common inflammatory rheumatic diseases.
comparison of the cytokine environment | day 1
  comparison cytokine environment within synovial biopsies from arthritis/bursitis occurring in the context of rare autoimmune/inflammatory syndromes or drug toxicity, n with that of arthritis/bursitis arising in common inflammatory rheumatic diseases.
Study of the gene expression profile of immune cells | day 1
  Study of the gene expression profile of immune cells present within synovial biopsies from arthritis/bursitis occurring in the context of rare autoimmune/inflammatory syndromes or drug toxicity,
Study of the gene expression profile of immune cells | day 1
  Study of the gene expression profile of immune cells present that of arthritis/bursitis occurring in common inflammatory rheumatic diseases."
comparison of the gene expression profile of immune cells | day 1
  comparison of the gene expression profile of immune cells in synovial biopsies from arthritis/bursitis occurring in the context of rare autoimmune/inflammatory syndromes or drug toxicity versus those from arthritis/bursitis occurring in common inflammatory rheumatic diseases

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU bordeaux, Bordeaux
  - CHU Brest - Hôpital Morvan, Brest

IPD SHARING:
Plan to Share IPD: Undecided